CLINICAL TRIAL: NCT00552019
Title: Inflammatory Changes of Corneal Thickness and Influence on Assessment of Intraocular Pressure
Brief Title: Intraocular Pressure (IOP) Assessed by Dynamic Contour Tonometer (DCT) and Goldman Applanation Tonometry (GAT)
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Responsible Party: Department of Ophthalmology at St. Franziskus Hospital, Department of Ophthalmology at St. Franziskus Hospital
Other Study IDs: 2007-405-f-S
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Uveitis; Intraocular Pressure
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate an assessment of the intraocular pressure with the dynamic contour tonometry and the Goldmann applanation tonometry in patients with active anterior uveitis.

DETAILED DESCRIPTION:
Keratoprecipitates are often found in anterior uveitis. Also elevation of the IOP can be seen in these patients. Goldmann applanation tonometry is the standard technique to assess the IOP but depends on the corneal thickness. Therefore IOP is measured by Goldmann and dynamic contour tonometry and corneal thickness is quantified by Orbscan at active uveitis and after the keratoprecipitates have disappeared.

ELIGIBILITY:
Inclusion Criteria:

* active anterior or panuveitis with keratoprecipitates

Exclusion Criteria:

* corneal endothelial dystrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary referral center
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
IOP by GAT and DCT | 3 months after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Heiligenhaus, MD, Study Director — Department of Ophthalmology at St.-Franziskus Hospital
Locations (1):
- Department of Ophthalmology at St.-Franziskus Hospital, Münster, Germany

REFERENCES:
- See also: Related Info — http://www.uveitis-zentrum.de